CLINICAL TRIAL: NCT01649466
Title: A Randomized Open-label Study to Compare Safety and Efficacy of Vildagliptin Versus NPH Insulin add-on to Glimepiride in Patients With Type 2 Diabetes Mellitus That do Not Reach Adequate Glycemic Control on Their Current Sulfonylurea Monotherapy.
Brief Title: Safety and Efficacy of Vildagliptin Versus NPH Insulin add-on to Glimepiride in Type 2 Diabetes Mellitus Patients.
Acronym: BENEFIT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237ADE08; 2012-001143-46 (EudraCT Number)
Record Dates: First submitted 2012-07-20; First posted 2012-07-25 (Estimated); Last update posted 2016-11-17 (Estimated); Status verified 2016-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus, diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — 1-(((3-hydroxy-1-adamantyl)amino)acetyl)-2-cyanopyrrolidine; Insulin

ARMS (2):
- Vildagliptin (Experimental): Patients randomized to the vildagliptin group will receive 50mg vildagliptin once daily add-on to their current glimepiride monotherapy for 24 weeks. No dose titrations are permitted during the study.
  Interventions: Drug: LAF237
- Protaphane (Active Comparator): Patients randomized to the Protaphane group will receive a individualized dose of Protaphane once daily as bedtime dose. The Protaphane dose will be titrated within the first 4 weeks to reach fasting plasma glucose values below 100 mg/dl.
  Interventions: Drug: Protaphane

INTERVENTIONS:
Drug: LAF237 — Vildagliptin will be used as commercially available tablets of 50mg.
  Arms: Vildagliptin
Drug: Protaphane — Protaphane will be used as commercially available injection pens
  Arms: Protaphane

SUMMARY:
This study is designed to evaluate safety and efficacy of vildagliptin versus NPH insulin add-on to glimepiride in patients with type 2 diabetes mellitus that do not reach adequate glycemic control on their current sulfonylurea monotherapy to give treating physicians a guidance which additional anti-diabetic treatment can be used if sulfonylurea monotherapy is not sufficient to reach glycemic control.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of type 2 diabetes mellitus.
* Contraindicated or intolerant to take metformin.
* HbA1c of ≥ 7.0% and ≤ 8.5%
* Current sulfonylurea (glimepiride) monotherapy and judged by the investigator to be inadequately controlled
* Other protocol-defined inclusion/exclusion criteria may apply

Exclusion Criteria:

* Patients who are taking any other anti-diabetes drug (oral or injection) other than an SU component in the preceding 12 weeks.
* Acute metabolic conditions such a ketoacidosis, lactic acidosis or hyperosmolar state within the past 6 month
* Patients taking sulfonylurea for longer than 5 years
* History of hypersensitivity to any of the study drugs or to drugs with similar chemical structures
* pregnancy
* Other protocol-defined inclusion/exclusion criteria may apply

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 162 (Actual)
Dates: Start 2012-08; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Percentage of patients reaching HbA1c below 7.0% without confirmed hypoglycemia and weight gain | 24 weeks
  Primary endpoint is proportion of patients reaching the combined endpoint, defined as a blood glucose target (HbA1c below 7.0%) without any confirmed hypoglycemic events (BG measurement < 3.9mM (71mg/dL)) and weight gain.
Rate of confirmed hypoglycemic events | 24 weeks
  Co-primary endpoint is to evaluate the rate of confirmed hypoglycemic events (BG measurement < 3.9mM (71mg/dL)) in type 2 diabetes patients treated with vildagliptin versus NPH insulin add-on to glimepiride.

SECONDARY OUTCOMES:
Incidence of severe hypoglycemic events | 24 weeks
  To evaluate the incidence of severe hypoglycemic events (suspected grade 2 and confirmed grade 2 events) in patients treated with vildagliptin versus NPH insulin add-on to glimepiride.
Incidence of symptomatic hypoglycemic events | 24 weeks
  To evaluate the incidence of symptomatic hypoglycemic events in patients treated with vildagliptin versus NPH insulin add-on to glimepiride.
Percentage of patients who reach their blood glucose target (HbA1c below 7.0%) without any confirmed hypoglycemic event | 24 weeks
  To evaluate the percentage of patients treated with vildagliptin versus NPH insulin add-on to glimepiride who reach their blood glucose target (HbA1c below 7.0%) without any confirmed hypoglycemic events.
Change from baseline in body weight at 24 weeks | Baseline, 24 week
  To evaluate body weight changes between study begin and study end in patients treated with vildagliptin versus NPH insulin add-on to glimepiride.
Change from baseline in HbA1c at 24 weeks | Baseline, 24 week
  To evaluate changes in HbA1c between study begin and study end in patients treated with vildagliptin versus NPH insulin add-on to glimepiride.
Change from baseline in Treatment Satisfaction Questionnaire for Medication (TSQM-9) at 24 week | Baseline, 24 week
  The TSQM-9 is a psychometrically sound and valid measure of the major dimensions of patients' satisfaction with medication.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (44):
- Germany (44):
  - Novartis Investigative Site, Anderbeck
  - Novartis Investigative Site, Augsburg
  - Novartis Investigative Site, Bad Kreuznach
  - Novartis Investigative Site, Bad Oeynhausen
  - Novartis Investigative Site, Balingen
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Cologne
  - Novartis Investigative Site, Dortmund
  - Novartis Investigative Site, Dresden
  - Novartis Investigative Site, Einbeck
  - Novartis Investigative Site, Eisleben Lutherstadt
  - Novartis Investigative Site, Elsterwerda
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Fulda
  - Novartis Investigative Site, Gelnhausen
  - Novartis Investigative Site, Graben-Neudorf
  - Novartis Investigative Site, Grossheirath-Rossach
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Hildesheim
  - Novartis Investigative Site, Kassel
  - Novartis Investigative Site, Kleve
  - Novartis Investigative Site, Lienen
  - Novartis Investigative Site, Löhne
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Mainz
  - Novartis Investigative Site, Mayen
  - Novartis Investigative Site, Mülheim
  - Novartis Investigative Site, München
  - Novartis Investigative Site, Oschatz
  - Novartis Investigative Site, Potsdam
  - Novartis Investigative Site, Reinfeld
  - Novartis Investigative Site, Saarlouis
  - Novartis Investigative Site, Saint Ingbert - Oberwuerzbach
  - Novartis Investigative Site, Schliemannstadt Neubukow
  - Novartis Investigative Site, Straubing
  - Novartis Investigative Site, Stuttgart
  - Novartis Investigative Site, Villingen-Schwenningen
  - Novartis Investigative Site, Wallerfing
  - Novartis Investigative Site, Wangen
  - Novartis Investigative Site, Wedemark
  - Novartis Investigative Site, Weiskirchen
  - Novartis Investigative Site, Wetzlar-Naunheim
  - Novartis Investigative Site, Wurzen
  - Novartis Investigative Site, Würzburg

REFERENCES:
- [Result] Forst T, Koch C, Dworak M. Vildagliptin versus insulin in patients with type 2 diabetes mellitus inadequately controlled with sulfonylurea: results from a randomized, 24 week study. Curr Med Res Opin. 2015 Jun;31(6):1079-84. doi: 10.1185/03007995.2015.1039936. Epub 2015 May 20. PMID 25867771
- [Result] Zuckermann A, Wang SS, Ross H, Frigerio M, Eisen HJ, Bara C, Hoefer D, Cotrufo M, Dong G, Junge G, Keogh AM. Efficacy and Safety of Low-Dose Cyclosporine with Everolimus and Steroids in de novo Heart Transplant Patients: A Multicentre, Randomized Trial. J Transplant. 2011;2011:535983. doi: 10.1155/2011/535983. Epub 2011 Sep 13. PMID 22295178